CLINICAL TRIAL: NCT05396404
Title: Using Empirical Mode Decomposition and Decision Tree to Extract the Balance and Gait Features and Classification in Sarcopenia
Brief Title: Empirical Mode Decomposition and Decision Tree in Sarcopenia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CCH IRB 211235
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-02

CONDITIONS: Sarcopenia; Fall; Gait, Unsteady; Balance; Distorted
Keywords: empirical mode decomposition; machine learning; decision tree
MeSH Terms: conditions — Sarcopenia; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation: all subject data were retrieved from databank which is stored in the e-medical chart system.

SUMMARY:
Sarcopenia is quickly becoming a major global public health issue. Falls are the leading cause of mortality among the elderly, and they must be addressed. The investigators will use machine learning techniques such as empirical mode decomposition technology and decision tree algorithms to extract the characteristics and classification of sarcopenia in this retrospective study in order to offer clinically proven and effective interventional strategies to prevent, stabilize, and reverse sarcopenia.

DETAILED DESCRIPTION:
Sarcopenia is becoming a severe global public health concern as the world's elderly population grows. Sarcopenia is characterized by muscular mass and strength loss, as well as impaired physical performance, and it is frequently connected with negative health outcomes such as falls. Falls are a primary cause of death in older individuals and must be addressed. Sarcopenia is currently diagnosed clinically using three primary technologies: imaging technology, precision medicine, and machine learning. In this study, the investigators will use previously collected data from nearly 200 community-dwelling subjects, including medical history, biochemistry, body composition, balance and gait, electromyography, and functional performance, to extract the characteristics and classification of sarcopenia using machine learning techniques such as empirical mode decomposition technology and decision tree algorithms. The investigators intend to offer clinically proven and effective interventional strategies to prevent, stabilize, and reverse sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* aged from 40 - 90
* DXA test performed
* blood sample tests were performed

Exclusion Criteria:

* stroke history
* amputation
* cancer related disease

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject's data were collected from the e-medical chart system.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
center of pressure (COP) | baseline: subject was enrolled
  Use computerized dynography to measure the postural sway displacement, velocity (etc., mm, mm/sec)
walking speed | baseline: subject was enrolled
  6m, patients can walk with foot orthosis and assistive devices
grip force | baseline: subject was enrolled
  Use a grip force meter (kg) to test both hands for test 3 times
step time | baseline: subject was enrolled
  Use computerized dynography to measure spatial gait parameter: step time (ms)
stance time | baseline: subject was enrolled
  Use computerized dynography to measure spatial gait parameter: stance time (ms)
swing time | baseline: subject was enrolled
  Use computerized dynography to measure spatial gait parameter: swing time (ms)
step / stance length | baseline: subject was enrolled
  Use computerized dynography to measure spatial gait parameter: step / stance distance (mm)
muscle thickness | baseline: subject was enrolled
  Use ultrasound to assess muscles morphological parameter: thickness (mm). Target muscles include quadriceps, hamstring, anterior tibialis, gastrocnemius.
international Quality of Life Assessment Short Form -36 (SF-36) | baseline: subject was enrolled
  including 8 health concepts: (1) physical functioning, (2) role limitations because of physical health problems; (3) bodily pain, (4) social functioning, (5) general mental health (psychological distress and psychological wellbeing), (6) role limitations because of emotional problems, (7) vitality (energy/fatigue), (8) general health perceptions.
  Scoring: answers to each question are scored which are then summed and transformed to a 0 - 100 scale.
  The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
amplitude of Muscle activity | baseline: subject was enrolled
  use electromyography to measure the muscles activity in microvolts (uv) included quadriceps, hamstrings, tibialis anterior, gastrocnemius during subject walking in self-selected speed in 6 meters.
Fear of fall scale | baseline: subject was enrolled
  A 15-item self-report questionnaire for measuring fear of falling. Each item is rated on a Likert-type scale from 1 (strongly disagree) to 4 (strongly agree). The total possible score ranges from 15-60, with higher scores indicating greater fear of falling.
Bone density | baseline: subject was enrolled
  A bone density test, DEXA, measures the mineral content of the bones in certain areas of the skeleton. A DEXA scan is a type of medical imaging test. It uses very low levels of x-rays to measure how dense participants' bones are. DEXA stands for "dual-energy X-ray absorptiometry." The bone density area includes: Hip and Spine
Body composition | baseline: subject was enrolled
  Dual energy x-ray absorptiometry (DEXA) measures bone mineral content (BMC), fat-free mass (FFM).

SECONDARY OUTCOMES:
concentration of CRP (C-Reactive Protein) | baseline: subject was enrolled
  The concentration of CRP in the blood test. CRP is used mainly as a marker of inflammation.
concentration of ALB (Serum albumin) | baseline: subject was enrolled
  The concentration of ALB in the blood test. Albumin is the most important contributor to the maintenance of plasma colloid oncotic pressure; deficiency results in edema.
concentration of Glomerular Filtration Rate (GFR) | baseline: subject was enrolled
  The concentration of GFR in the blood test. The glomerular filtration rate is the best test to measure the patient's level of kidney function and determine the stage of kidney disease. It can calculate it from the results of the blood creatinine test.
concentration of Hemoglobin (Hb) | baseline: subject was enrolled
  The concentration of Hb in the blood test.
concentration of Glucose SPOT | baseline: subject was enrolled
  The concentration of Glucose SPOT in the blood test. TheSpot glucose measurement in epidermal interstitial fluid appears to be a promising alternative to capillary blood glucose estimation
concentration of Cholesterol | baseline: subject was enrolled
  The concentration of Cholesterol in the blood test.
concentration of Triglyceride | baseline: subject was enrolled
  The concentration of Triglyceride in the blood test.
concentration of Transferrin | baseline: subject was enrolled
  The concentration of Transferrin in the blood test.
Berg balance test (BBS) | baseline: subject was enrolled
  including 14 items which are scored on a 5 points scale (0-4). The degree of success in achieving each task is given a score of zero (unable) to four (independent), and the final measure is the sum of all of the scores.
  The item scores are summed, minimum score =0, maximum score = 56
Body Mass Index (BMI) | baseline: subject was enrolled
  (body weight) kg/(height) m*(height)m
Mini-mental state examination (MMSE) | baseline: subject was enrolled
  It is an 11-question measure that tests five areas of cognitive function:
  orientation, registration, attention and calculation, recall, and language. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment.
calf muscle circumference | baseline: subject was enrolled
  Use ruler to measure the bilateral calf muscle circumference, It is an anthropometric parameter commonly used in clinical practice.
Timed up and go | baseline: subject was enrolled
  To determine fall risk and measure the progress of balance, sit to stand and walking. Patients wear their regular footwear and can use a walking aid, if needed. The patient starts in a seated position. The patient stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated. To document if the assistive device used. Stopwatch to record the whole task duration.

CONTACTS AND LOCATIONS:
Overall Officials: TASEN WEI, MD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan